CLINICAL TRIAL: NCT06725849
Title: Barriers to Physical Activity and Exercise in Patients With Familial Mediterranean Fever
Brief Title: Barriers to Physical Activity in Familial Mediterranean Fever
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Tugba Civi Karaaslan, PhD., Istanbul University - Cerrahpasa
Other Study IDs: ISTANBULC6
Record Dates: First submitted 2024-10-17; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Familial Mediterranean Fever (FMF )
Keywords: exercise; Physical Activity
MeSH Terms: conditions — Familial Mediterranean Fever; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project is a 2209-A TÜBİTAK project. It has been developed to identify the barriers to physical activity among patients diagnosed with Familial Mediterranean Fever (FMF).

The project aims to determine the problems encountered by FMF patients when engaging in physical activity and the reasons behind these issues, using various assessment methods to identify the reasons for avoiding physical activity.

DETAILED DESCRIPTION:
This project is a 2209-A TÜBİTAK project. It has been developed to identify the barriers to physical activity among patients diagnosed with Familial Mediterranean Fever (FMF) referred to the Department of Internal Medicine, Rheumatology Division, at Istanbul University-Cerrahpaşa, Cerrahpaşa Medical Faculty, as well as the Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation.

The project aims to determine the problems encountered by FMF patients when engaging in physical activity and the reasons behind these issues, using various assessment methods to identify the reasons for avoiding physical activity. Patients diagnosed with FMF will be evaluated based on pain (McGill Melzack Pain Questionnaire), quality of life (FMF Quality of Life Measure), fatigue status (Fatigue Severity Scale), kinesiophobia (Tampa Scale for Kinesiophobia), grip strength (Digital Hydraulic Hand Dynamometer), and aerobic capacity (Spirometer).

Assessments will be conducted twice a week for three months, with each session lasting 30 minutes, utilizing the Digital Hydraulic Hand Dynamometer and Spirometer under the supervision of researchers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Familial Mediterranean Fever (FMF)
* Ability to respond to the questionnaires
* Capability to engage in physical activity

Exclusion Criteria:

* Any form of disability (visual, auditory, mental, physical)
* Illiteracy in Turkish
* Presence of comorbidities that may hinder assessment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Familial Mediterranean Fever (FMF) referred to the Department of Internal Medicine, Rheumatology Division, at Istanbul University-Cerrahpaşa, Cerrahpaşa Medical Faculty, as well as the Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-16 (Estimated); Primary Completion 2025-12-16 (Estimated); Study Completion 2025-12-16 (Estimated)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire Short | It will be applied once for up to 6 months.
  Prepared with the support of the World Health Organization (WHO) and the Centers for Disease Control and Prevention (CDC), this standardized questionnaire has been developed by researchers from different countries. The questionnaire has both long and short forms. We will evaluate our participants using the short form consisting of 7 items. Sağlam et al. have conducted validity and reliability studies for the Turkish version of the questionnaire. The survey inquires about the time spent on physical activities over the past 7 days. It consists of 7 questions. Questions 1 and 2 ask about the time spent on vigorous physical activities, specifically how many days per week and how many minutes (or hours) per day. Questions 3 and 4 focus on moderate-intensity activities, while questions 5 and 6 inquire about the time spent walking, asking how many days per week and how many minutes (or hours) per day. The last question asks about the time spent sitting, inquiring how many minutes (or hours).
Familial Mediterranean Fever Quality of Life Scale | It will be applied once for up to 6 months.
  Developed with the support of the World Health Organization (WHO) and the Centers for Disease Control and Prevention (CDC) by researchers from different countries, the scale consists of 20 questions and is based on four factors, developed using psychometric methods. The factor groups represent four different dimensions related to quality of life in Familial Mediterranean Fever. Factor 1 is associated with physical impact, Factor 2 with social and recreational impact, Factor 3 with psychological impact, and Factor 4 with the impact of sleep.The FMF Quality of Life (FMF QL) scale has a strong relationship with other generic quality of life questionnaires (such as SF-36 and EUROHIS) and a moderate relationship with disability, sleep, and depression scales that may be related to quality of life. The relationships of the questionnaire with parameters not directly related to quality of life are weak to moderate or nonsensical, which demonstrates the distinctive feature of our questionnaire.

SECONDARY OUTCOMES:
McGill Melzack Pain Questionnaire | It will be applied once for up to 6 months.
  Developed by Melzack and Targerson in 1971, the questionnaire has undergone validity and reliability studies in Turkish by Eti Aslan and Olgun. The questionnaire consists of four subsections. The introductory section inquires about the patient's name, age, medical diagnosis/issues, the type and dosage of analgesics used, and the patient's level of cognition.
  The first section asks about the location and type of pain (deep - D / superficial - Y). The second section asks the individual to describe their current pain. The third section examines the relationship of pain with time, consisting of three questions aimed at determining the continuity, frequency, and factors that increase or decrease the pain.
  The fourth section assesses the intensity of the pain, with five word groups ranging from mild to unbearable. The total score ranges from 0 to 112.
Tampa Scale for Kinesiophobia-Fatigue | It will be applied once for up to 6 months.
  The original Tampa Scale for Kinesiophobia (TSK) was developed by Miller, Kopri, and Todd in 1991 but was not published. Vlaeyen and colleagues re-published the original scale, consisting of 17 items, in 1995 with the permission of the original developers. The TSK is a 17-item questionnaire designed to measure fear of movement/re-injury. The scale includes parameters related to work-related activities, injury/re-injury, and fear-avoidance.
  Vlaeyen and colleagues later created two shorter forms of this scale, each consisting of 13 items. Fear of movement is a significant issue that negatively impacts patients' quality of life, leading to varying degrees of disability and participation problems. It is essential to identify this issue and consider the patients' fears of movement in addition to implementing targeted treatments in treatment programs.
Fatigue Severity Scale | It will be applied once for up to 6 months.
  The scale consists of 9 questions, each with a score ranging from 1 to 7. An increase in the scale score indicates a higher level of fatigue. In 2007, Armutlu and colleagues conducted validity and reliability studies for the scale in Turkey. The scale assesses individuals' fatigue levels over the past month, as studied by Yorulmaz et al. in patients with sleep apnea.
  Responses are scored from "Not at all agree (1)" to "Completely agree (7)." The scale score is the average value of the responses. If the average score is 5 or higher, it is evaluated as "fatigue present.
Digital Hydraulic Hand Dynamometer | It will be applied once for up to 6 months.
  Hydraulic devices that use kilograms or pounds as measurement units allow for the measurement of static grip strength. A digital hydraulic hand dynamometer will be used to measure the participants' gross grip strength. Gross grip refers to the grasping motion used to hold an object in the palm of the hand.
  During the measurement, the hand is in a pinch grip position, and the metacarpophalangeal joints are in a flexed position. The gripping section of the device can be adjusted to different levels according to the size of the hand. The patient sits in a chair with the shoulder in a neutral position, the elbow flexed at 90 degrees, the forearm resting on the table, and the wrist in a neutral position. The participant is instructed to perform a strong grip.
  The measurement is repeated three times, and the average of the three values is recorded in kilograms.
Aerobic Capacity Assessment: Spirometer | It will be applied once for up to 6 months.
  A spirometer is a device used to measure respiratory function.Currently, flow meters are commonly used. The sensors in the device are sensitive to flow, and they calculate volume based on the measured flow. The values provided for the patient are compared to reference data.Flow-type spirometers are easy to clean and disinfect, and the devices must be calibrated daily.The test is performed in a seated position. A clip is placed on the patient's nose, and they are instructed to take a disposable mouthpiece and hold it tightly with their lips. The individual is asked to breathe in and out 4 to 5 times at normal tidal volume through the spirometer mouthpiece. Then, they are instructed to take a deep breath and exhale quickly and forcefully. The exhalation should be continuous for at least 6 seconds. After sufficient exhalation, the individual is instructed to take a deep breath to conclude the test. The test is repeated three times, and the highest value is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)